CLINICAL TRIAL: NCT00658567
Title: A Study of Safety and Efficacy of Pimavanserin (ACP-103) in Patients With Parkinson's Disease Psychosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-014
Record Dates: First submitted 2008-04-10; First posted 2008-04-15 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Parkinson's Disease Psychosis
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2 (Experimental): pimavanserin tartrate (ACP-103) 20 mg, tablet, once daily by mouth, 6 weeks
  Interventions: Drug: Pimavanserin tartrate (ACP-103)
- Placebo (Placebo Comparator): Placebo tablet, once daily by mouth, 6 weeks
  Interventions: Drug: Pimavanserin tartrate (ACP-103)
- 1 (Experimental): pimavanserin tartrate (ACP-103) 10 mg, tablet, once daily by mouth, 6 weeks
  Interventions: Drug: Pimavanserin tartrate (ACP-103)

INTERVENTIONS:
Drug: Pimavanserin tartrate (ACP-103) — 10 mg, tablet, once daily by mouth, for six weeks
  Arms: 1
Drug: Pimavanserin tartrate (ACP-103) — 20 mg, tablet, once daily by mouth, for six weeks
  Arms: 2
Drug: Pimavanserin tartrate (ACP-103) — Placebo, tablet, once daily by mouth, for six weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of two dose levels of pimavanserin (ACP-103) compared to placebo in patients with Parkinson's disease psychosis.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Parkinson's disease with a minimum duration of 1 year
* Presence of visual and/or auditory hallucinations, and/or delusions, occurring during the four weeks prior to study screening
* Psychotic symptoms must have developed after Parkinson's disease diagnosis was established
* Subject must be on stable dose of anti-Parkinson's medication for 1 month prior to Study Day 1 (Baseline) and during the trial
* Subject that has received stereotaxic surgery for subthalamic nucleus deep brain stimulation must be at least 6 months post surgery and the stimulator settings must have been stable for at least 1 month prior to Study Day 1 (Baseline) and must remain stable during the trial
* The subject is willing and able to provide consent
* Caregiver is willing and able to accompany the subject to all visits

Exclusion Criteria:

* Subject has a history of significant psychotic disorders prior to or concomitantly with the diagnosis of Parkinson's disease including, but not limited to, schizophrenia or bipolar disorder
* Subject has received previous ablative stereotaxic surgery (i.e., pallidotomy and thalamotomy) to treat Parkinson's disease
* Subject has current evidence of a serious and or unstable cardiovascular, respiratory, gastrointestinal, renal, hematologic or other medical disorder
* Subject has had a myocardial infarction in last six months
* Subject has any surgery planned during the screening, treatment or follow-up periods

Patients will be evaluated at screening to ensure that all criteria for study participation are met. These evaluations will include specific measures of psychosis severity, delirium, dementia, cardiovascular condition, and pregnancy status. Patients may be excluded from the study based on these assessments (and specifically if it is determined that their baseline health and psychiatric condition do not meet all protocol-specified entry criteria).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (25):
  - La Habra, California
  - Laguna Hills, California
  - Reseda, California
  - Ventura, California
  - Englewood, Colorado
  - Farmington, Connecticut
  - Deerfield Beach, Florida
  - Panama City, Florida
  - Sarasota, Florida
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Clinton, Michigan
  - Detroit, Michigan
  - East Lansing, Michigan
  - Columbia, Missouri
  - Omaha, Nebraska
  - Albany, New York
  - Commack, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - New Bern, North Carolina
  - Toledo, Ohio
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Burlington, Vermont
- Innsbruck, Austria
- Belgium (3):
  - Brussels
  - Ottignies
  - Roeselare
- Italy (3):
  - Chieti Scalo
  - Grossetto
  - Roma
- Poland (4):
  - Bydgoszcz
  - Katowice
  - Lodz
  - Lublin
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Belgrade, Serbia
- Spain (3):
  - Barcelona
  - Donostia / San Sebastian
  - Santiago de Compostela
- Sweden (3):
  - Jönköping
  - Linköping
  - Stockholm

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimavanserin 10 mg: Pimavanserin tartrate (ACP-103) 10 mg, tablet, once daily by mouth, 6 weeks
- Pimavanserin 20 mg: Pimavanserin tartrate (ACP-103) 20 mg, tablet, once daily by mouth, 6 weeks
Period: Overall Study
Arm/Group | Placebo | Pimavanserin 10 mg | Pimavanserin 20 mg
Started | 40 | 42 | 41
Completed | 32 | 38 | 35
Not Completed | 8 | 4 | 6
Not completed — Adverse Event | 5 | 2 | 3
Not completed — Voluntary Withdrawal of Consent | 2 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — At Discretion of Sponsor | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- 10 mg: Pimavanserin tartrate (ACP-103) 10 mg, tablet, once daily by mouth, 6 weeks
- 20 mg: Pimavanserin tartrate (ACP-103) 20 mg, tablet, once daily by mouth, 6 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg | 20 mg | Total
Number analyzed (Participants) | 39 | 41 | 41 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 7 | 21
  >=65 years | 32 | 34 | 34 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (7.91) | 71.0 (7.44) | 72.1 (8.15) | 72.0 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 17 | 44
  Male | 27 | 26 | 24 | 77
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 18 | 53
  Europe | 21 | 24 | 23 | 68

OUTCOME MEASURES:

1. Primary Outcome: Antipsychotic Efficacy
Description: Antipsychotic efficacy was defined as a decrease in the severity and/or frequency of hallucinations and/or delusions. This is measured as the change from baseline (Day 1) to Day 42 in the Scale for the Assessment of Positive Symptoms - Hallucinations and Delusions scales (SAPS-H+D) score for the ITT Analysis Set. The possible total score is 1 to 100 and a negative change in score indicates improvement.
  Analysis Method: Analysis of Covariance (ANCOVA) and missing data was imputed using Last Observation Carried Forward (LOCF) method.
Time Frame: Each study visit (i.e. Days 1, 8, 15, 29 and 42)
Population: This is the "Intent to Treat" population, defined as patients who received at least one dose of study drug and had both the baseline SAPS assessment and at least one post-baseline SAPS assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on the SAPS H+D scale
Arm/Group | Placebo | Pimavanserin 10 mg | Pimavanserin 20 mg
Number analyzed (Participants) | 38 | 38 | 41
Scores on the SAPS H+D scale
  Change from Baseline | -4.4 [-6.5 to -2.3] | NA [NA to NA] — Only the high dose comparison was incorporated in the ANCOVA model analysis following the early termination of the study. The prospective SAP eliminated the analysis of the low dose, 10 mg arm. | -6.5 [-8.5 to -4.5]
  Difference of Least Squares Mean versus Placebo | NA [NA to NA] — Calculation is a comparison of active arm versus placebo. | NA [NA to NA] — Only the high dose comparison was incorporated in the ANCOVA model analysis following the early termination of the study. The prospective SAP eliminated the analysis of the low dose, 10 mg arm. | -2.1 [-4.9 to 0.8]

2. Secondary Outcome: Motor Symptoms Change From Baseline (Negative = Improvement)
Description: Motor symptoms were measured using the change from baseline (Day 1) to Day 42 in the combined score of the Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living) and Part III (Motor Examination). The total possible score is 0 to 160 and a negative change in score indicates improvement.
  Analysis Method: ANCOVA, and missing data was imputed using LOCF method. The UPDRS Parts II+III score was analyzed by constructing 2-sided 95% confidence intervals (CIs) on the difference between each pimavanserin dose group and placebo mean change from baseline. Non-inferiority was concluded if the upper limit of the CI was less than or equal to 5.
Time Frame: Each study visit (i.e. Days 1, 8, 15, 29 and 42)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on UPDRS-II+III scale.
Arm/Group | Placebo | Pimavanserin 10 mg | Pimavanserin 20 mg
Number analyzed (Participants) | 38 | 38 | 41
Score on UPDRS-II+III scale.
  Change from Baseline | -1.8 [-4.6 to 1.0] | NA [NA to NA] — Only the high dose comparison was incorporated in the ANCOVA model analysis following the early termination of the study. The prospective SAP eliminated the analysis of the low dose, 10 mg arm. | -3.9 [-6.6 to -1.2]
  Difference of Least Squares Mean versus Placebo | NA [NA to NA] — Calculation is a comparison of active arm versus placebo. | NA [NA to NA] — Only the high dose comparison was incorporated in the ANCOVA model analysis following the early termination of the study. The prospective SAP eliminated the analysis of the low dose, 10 mg arm. | -2.1 [-5.9 to 1.8]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: From the time the informed consent was signed, adverse events were recorded in the subject's source documents and entered into the appropriate eCRF pages at the Screening visit, at visits on Study Days 1, 8, 15, 29, 42 and Day 70 or 4 weeks after the last dose for subjects who do not continue into the open-label, extension protocol.
Arm/Group | Placebo | Pimavanserin 10 mg | Pimavanserin 20 mg
Serious Adverse Events (participants affected / at risk) | 2/39 | 3/41 | 1/41
Other Adverse Events (participants affected / at risk) | 12/39 | 4/41 | 8/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=39) | Pimavanserin 10 mg (N=41) | Pimavanserin 20 mg (N=41)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Delusional disorder, persecutory type (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=39) | Pimavanserin 10 mg (N=41) | Pimavanserin 20 mg (N=41)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 2 (3) | 3 (3)
Hallucination (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.